CLINICAL TRIAL: NCT02859623
Title: Descriptive Study of the Efficacy of Treatments for Blastic Dendritic Cell Neoplasm (BPDCN): a Retrospective Study of Patients Diagnosed in France From 2000 to 2013
Brief Title: Descriptive Study of the Efficacy of Treatments for Blastic Dendritic Cell Neoplasm (BPDCN)
Acronym: LpDC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: LpDC
Record Dates: First submitted 2016-07-21; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm; Hematological Malignancies
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; Hematologic Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Blastic plasmacytoid dendritic cell neoplasm (BPDCN) is a rare disease characterized by an aggressive clinical behavior and a poor prognosis. It predominantly affects elderly males with an average age of 67 years at diagnosis and the affected organs are usually the skin, bone marrow, lymph nodes and the central nervous system. Patients with BPDCN have poor outcomes with median overall survival (OS) ranging in the largest series of patients from 8 to 12 months.

Patient care must be defined in this pathology. Despite 40%-90% complete remission (CR) rates after initial chemotherapy, relapses are almost inevitable.

The investigators have developed a national network to collect clinical and biological data of French patients diagnosed with BPDCN.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with blastic plasmacytoid dendritic cell neoplasm (BPDCN) from January 2000 to June 2013 in France.
* Diagnosis should be established by hematology laboratory of French blood Agency of Bourgogne Franche-Comté and/or by anatomopathological analysis (realized in local centres or by Tony Petrella at Dijon University Hospital) according to phenotypic and anatomopathological criteria published in the literature.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study concerns patients diagnosed with blastic plasmacytoid dendritic cell neoplasm (BPDCN) from January 2000 to June 2013.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
description of the efficacy of treatments for BPDCN | from the diagnosis to death or until June 2013, date of end of data collection
  Measurement of the overall survival for all patients from the date of diagnostic until death or end of data collection

SECONDARY OUTCOMES:
description of clinical profiles of patients | from the diagnosis to death or until June 2013, end of data collection
  presence of cutaneous lesions
description of biological profiles of patients | from the diagnosis to death or until June 2013, end of data collection
  immunophenotyping profile
complete remission rate | from the diagnosis to death or until June 2013, end of data collection
mean duration of the first remission | from the diagnosis to death or until June 2013, end of data collection
survival without events | from the diagnosis to death or until June 2013, end of data collection
non-responders rate | from the diagnosis to death or until June 2013, end of data collection
time interval between two treatments | from the diagnosis to death or until June 2013, end of data collection
mortality without relapse | from the diagnosis to death or until June 2013, end of data collection